CLINICAL TRIAL: NCT00773929
Title: A Multicenter Phase I Clinical and Pharmacokinetic Study of Oral TAK-593 in Subjects With Nonhematologic Advanced Cancer
Brief Title: Safety Study of TAK-593 Given Orally in Subjects With Nonhematologic Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Clinical Research Monitor, Millennium Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-593_101
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Solid Tumors
MeSH Terms: interventions — TAK 593

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 3-6 subjects each cohort. Escalate dose after safety evaluation of subjects in cohort
  Interventions: Drug: TAK-593

INTERVENTIONS:
Drug: TAK-593 — Tablets of TAK-593 investigational drug for oral administration, tablets in 2 strengths: 1 mg and 4 mg tablets.
  Administration will initially be 4 mg, once a day and transition to 2 mg BID schedule dependant on safety

SUMMARY:
The purpose of this study is to determine the safety and toxicity profile of TAK-593 and determine the maximum tolerated dose of TAK-593.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age diagnosed with advanced solid tumor cancer that failed to respond to standard therapies and where no other treatment options are available.
* No prior chemotherapy
* Able to understand and follow study requirements
* Subject or subject's legal representative signs a written, informed consent form prior to beginning any study procedures.
* Women who are post-menopausal for at least 1 year before screening or surgically sterile
* Women of childbearing potential agree to practice two effective methods of birth control from the time of signing the informed consent form through 30 days after the last dose of the study drug or agree to completely abstain from heterosexual intercourse.
* Men who agree to practice an effective method of birth control for the entire study treatment period and through 30 days after the last dose of study drug or completely agree to abstain from heterosexual intercourse.
* Ability to swallow and retain oral medication
* Meet study specific laboratory test standards for bone marrow function, liver function, blood pressure, and renal function.

Exclusion Criteria:

* Cancer has spread to the brain
* History of another cancer diagnosed or treated within the past 3 years.
* Severe cardiovascular issues including heart attack within the past 6 months, unstable angina or arrhythmias that require treatments.
* Severe thyroid disease
* Unstable angina
* Arrhythmia issues
* History of bleeding issues
* Serious wounds, ulcers or bone fractures that do not heal
* Subject is pregnant or breast feeding
* Subject has illnesses or conditions that may affect their ability to participate in the study
* Subject participated in another clinical study/post marketing clinical study within 4 weeks prior to the start of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Toxicities of TAK-593 Pharmacokinetic parameters of TAK-593 | 18-24 months

SECONDARY OUTCOMES:
Response outcomes including objective response and clinical benefit response. | 18-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States